CLINICAL TRIAL: NCT01646749
Title: Effects of Beef Protein Consumption on Energy Intake - The Protein Leverage Hypothesis
Brief Title: Effects of Beef Protein Consumption on Energy Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: National Cattlemen's Beef Association, a contractor to the Beef Checkoff (Industry)
Responsible Party: Principal Investigator, Eveline Martens, PhD student, Maastricht University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NL41371
Record Dates: First submitted 2012-07-16; First posted 2012-07-20 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Obesity; Severe Overweight
Keywords: Energy intake; Beef protein; Satiety; Protein leverage hypothesis
MeSH Terms: conditions — Obesity; Overweight | interventions — Meals

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Protein intake of 5 energy percent (En%) (Experimental)
  Interventions: Dietary Supplement: Differences in protein content (En%) of meals
- Protein intake of 15 En% (Experimental)
  Interventions: Dietary Supplement: Differences in protein content (En%) of meals
- Protein intake of 30 En% (Experimental)
  Interventions: Dietary Supplement: Differences in protein content (En%) of meals

INTERVENTIONS:
Dietary Supplement: Differences in protein content (En%) of meals — The three applied conditions will differ in the relative protein content of the meals, including 5 En%, 15 En% and 30 En% from protein. Beef protein will be used as main meat protein source in the 15 En% and 30 En% protein conditions. The resulting macronutrient compositions of the diets will be En% Protein/Carbohydrate/Fat; 5/60/35, 15/50/35, and 30/35/35. All meals (breakfast, lunch, dinner) within each condition will have the same macronutrient composition. All food items, and the energy density, weight and volume of the meals will be the same between conditions. All snack items will be very low in protein content.
  Other Names: All food items will be commercial available.

SUMMARY:
The purpose of this study is to determine ad libitum daily energy intake, body weight changes and appetite profile in response to protein/carbohydrate and fat ratio over 12 consecutive days, and in relation to age, gender, body mass index (BMI) and fat mass and obesity-associated (FTO) gene alleles.

DETAILED DESCRIPTION:
The protein leverage hypothesis requires specific evidence whether energy intake would depend on a possible protein intake target in humans. Meat protein as complete protein may show most beneficial effects on variables regarding food intake regulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Age 18-70 years
* BMI 18-35 kg/m2
* Non-smoking
* Weight stable

Exclusion Criteria:

* Smoking
* Use of medication
* More than moderate alcohol consumption
* Vegetarian

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Body weight change | 11 days
  Body weight will be measured on day 1, 6 and 12. Subsequently, the change in body weight over time will be calculated.
Appetite profile | 12 consecutive days
  Appetite profile will be measured by means of questionnaires: visual analogue scales (VAS). Area under the curve (AUC) will be calculated over 12 consecutive days.
Energy intake | 12 consecutive days
  Total energy intake over 12 days will be determined for each subject by adding energy intake during meals to energy intake from snack consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Margriet S Westerterp-Plantenga, Prof. dr., Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands

REFERENCES:
- [Background] Simpson SJ, Raubenheimer D. Obesity: the protein leverage hypothesis. Obes Rev. 2005 May;6(2):133-42. doi: 10.1111/j.1467-789X.2005.00178.x. PMID 15836464
- [Background] Weigle DS, Breen PA, Matthys CC, Callahan HS, Meeuws KE, Burden VR, Purnell JQ. A high-protein diet induces sustained reductions in appetite, ad libitum caloric intake, and body weight despite compensatory changes in diurnal plasma leptin and ghrelin concentrations. Am J Clin Nutr. 2005 Jul;82(1):41-8. doi: 10.1093/ajcn.82.1.41. PMID 16002798
- [Background] Griffioen-Roose S, Mars M, Siebelink E, Finlayson G, Tome D, de Graaf C. Protein status elicits compensatory changes in food intake and food preferences. Am J Clin Nutr. 2012 Jan;95(1):32-8. doi: 10.3945/ajcn.111.020503. Epub 2011 Dec 7. PMID 22158729
- [Background] Gosby AK, Conigrave AD, Lau NS, Iglesias MA, Hall RM, Jebb SA, Brand-Miller J, Caterson ID, Raubenheimer D, Simpson SJ. Testing protein leverage in lean humans: a randomised controlled experimental study. PLoS One. 2011;6(10):e25929. doi: 10.1371/journal.pone.0025929. Epub 2011 Oct 12. PMID 22022472
- [Background] Mikkelsen PB, Toubro S, Astrup A. Effect of fat-reduced diets on 24-h energy expenditure: comparisons between animal protein, vegetable protein, and carbohydrate. Am J Clin Nutr. 2000 Nov;72(5):1135-41. doi: 10.1093/ajcn/72.5.1135. PMID 11063440
- [Derived] Martens EA, Tan SY, Mattes RD, Westerterp-Plantenga MS. No protein intake compensation for insufficient indispensable amino acid intake with a low-protein diet for 12 days. Nutr Metab (Lond). 2014 Aug 20;11:38. doi: 10.1186/1743-7075-11-38. eCollection 2014. PMID 25183991
- [Derived] Martens EA, Tan SY, Dunlop MV, Mattes RD, Westerterp-Plantenga MS. Protein leverage effects of beef protein on energy intake in humans. Am J Clin Nutr. 2014 Jun;99(6):1397-406. doi: 10.3945/ajcn.113.078774. Epub 2014 Apr 23. PMID 24760974